CLINICAL TRIAL: NCT01467310
Title: Defining the Triple Negative Breast Cancer Kinome Response to GSK1120212
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry); National Cancer Institute (NCI) (NIH); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LCCC 1122; 11-1689 (Other: UNC IRB); CA058223 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2011-10-13; First posted 2011-11-08 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
Keywords: GSK1120212; TNBC; Triple Negative Breast Cancer; Surgical Resection
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GSK1120212 (Experimental)
  Interventions: Drug: GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — 1.5 to 2.0 mg taken orally every day for seven days.

SUMMARY:
Research into treatments for breast cancer relies more and more on an understanding of how the cells of tumor tissue act when they are exposed to a new or different drug. To find these new or different drugs to treat cancer, researchers are looking at proteins that help cancer cells grow, such as a group of proteins called Kinases. In this study the investigators want to look at the activity of kinases when a particular experimental drug called GSK1120212 is administered. GSK1120212 blocks a kinase called MEK. GSK1120212 is not yet approved by the FDA for use in breast cancer patients. The investigators want to give subjects GSK1120212 for a short period of time (one week) to see how MEK and the other kinases function in cancer cells both before and after the study drug is given. This study is not intended to treat cancer, it is looking at ways that the investigators may treat cancer in the future.

DETAILED DESCRIPTION:
In this study the investigators want to look at the activity of kinases when a particular experimental drug called GSK1120212 is administered. GSK1120212 blocks a kinase called MEK. GSK1120212 is not yet approved by the FDA for use in breast cancer patients. The investigators want to give subjects GSK1120212 for a short period of time (one week) to see how MEK and the other kinases function in cancer cells both before and after the study drug is given. The investigators are giving this drug for research purposes only. The length of time it is being given is not intended to treat cancer.

Research into treatments for breast cancer relies more and more on an understanding of how the cells of tumor tissue act when they are exposed to a new or different drug. To find these new or different drugs to treat cancer, researchers are looking at proteins that help cancer cells grow, such as a group of proteins called Kinases. This is important because many of the newest cancer drugs are designed to block kinases causing the cancer cells to die and the tumors to shrink. However, blocking only one of the kinases at a time is often less effective than the investigators expected because when you block one kinase another can take its place. For this reason, the investigators may need to treat breast cancer with more than one kinase-blocking drug at a time. However, the investigators don't yet know what the best combination of drugs should be, because it is hard to measure all the possible kinases. Previous studies have only been able to identify less than 10% of the hundreds of kinases in cancer cells.

Recently researchers here at UNC have developed a process that can identify may (more than half) of these kinases. This can tell us which kinases need to be blocked at the same time to make tumors shrink so that the investigators can design the best combinations of kinase blocking drugs for triple negative breast cancer. This is especially important for individuals with triple negative breast cancer (TNBC) because there are fewer drugs available that can block molecules that affect tumor growth. The investigators believe that kinase-blocking drugs have the potential to be a more effective treatment for people with TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed TNBC (i.e., ER negative, PR negative (each <10% staining by immunohistochemistry) and Her2 negative (0-1+ or FISH non-amplified; by clinical assay on primary tumor)
* Stage I-IIIc disease:

  * Scheduled for lumpectomy or mastectomy
  * No prior or current therapy for breast cancer
  * Not considered candidate for therapeutic neoadjuvant treatment
* For stage IV disease:

  * Scheduled for surgical resection of oligometastatic disease
  * Previously untreated for breast cancer
* Subject enrolls into LCCC9819
* ECOG Performance Status 0-2
* Normal end organ function as defined by the following:

  * Absolute neutrophil count (ANC)≥ 1.2 X 109/L;
  * Hemoglobin ≥ 9 g/dL;
  * Platelets ≥ 75 X 109/L;
  * PT/INR and PTT ≤ 1.2 X upper limit of normal (ULN);
  * Albumin ≥ 2.5 g/dL
  * Total bilirubin ≤ 1.5 x ULN mg/dL
  * AST and ALT ≤ 2.5 X ULN
  * Creatinine ≤ 1.5 X ULN OR Calculated creatinine clearance ≥50 mL/min OR 24-hour urine creatinine clearance ≥50 mL/min;
  * Ejection fraction ≥ LLN by ECHO (preferred) or MUGA
* Age ≥18 years
* Willing to use adequate contraception if applicable, and to continue use for 4 weeks post last dose of GSK1120212
* Sufficient fresh or frozen tissue remaining from pre-treatment core incisional biopsy or willing to undergo biopsy for research purposes only (approximately 10mg or one core's worth of tissue needed)
* Surgeon and Medical Oncologist agree one week window trial appropriate/safe for trial candidate and that surgery appointment can accommodate a 7 day (one week) treatment schedule
* Able to swallow oral medications

Exclusion Criteria

* Pregnant or lactating female
* Currently active GI disease, or prior surgery that may affect ability to absorb oral medications
* Prior radiation therapy to the target lesion
* History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR):

  * History of RVO or CSR, or predisposing factors to RVO or CSR (e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
* Current use of a prohibited medication or requires any of these medications during treatment with GSK1120212 (see section 4.6).
* Use of an investigational anti-cancer drug within 28 days or five half-lives, whichever is shorter, prior to the first dose of GSK1120212. A minimum of 10 days between termination of the investigational drug and administration of GSK1120212 is required. In addition, any drug-related toxicity should have recovered to Grade 1 or less.
* Prior treatment with MEK or BRAF inhibitors
* Any major radiotherapy, or immunotherapy within the last four weeks; use of erythropoietin replacement or bisphosphonates is considered supportive care and their use is permitted
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease)
* History or evidence of cardiovascular risk including any of the following:

  * QTc interval >/= 480 msecs.
  * Clinically significant uncontrolled arrhythmias Exception: subjects with controlled atrial fibrillation for >30 days prior to day 1 of treatment with GSK1120212 are eligible
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within the past 24 weeks
  * ≥Class II heart failure as defined by the New York Heart Association (NYHA) functional classification system (see Appendix C)
* Known human immunodeficiency virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection which will be allowed)
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug, dimethyl sulfoxide (DMSO), or excipients
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol
* Any other concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

PRIMARY OUTCOMES:
the number and type of kinases in participant tissue sample prior to administration of drug compared to post-treatment. | Two years
  use of pan kinase inhibitors immobilized on beads to capture expressed kinases in cells and tumors. The activation state of more than 60% of the expressed kinome, defined by RNA-seq, will be analyzed using mass spectrometry analysis of the captured kinases.

SECONDARY OUTCOMES:
the number and type of kinases that produce a compensatory response to MEK inhibitor | Two years
  The activation state of more than 60% of the expressed kinome, defined by RNA-seq, will be analyzed using mass spectrometry analysis of the captured kinases. For each activated kinase, a drug therapy that combines an inhibitor of that kinase with a MEK inhibitor will be identified.
the number of participants with adverse events | Two years
  Identify any safety issues in subjects treated with drug GSK1120212

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carey, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States